CLINICAL TRIAL: NCT02594722
Title: Metabolism and Oxygen Consumption During Functional Electrical Stimulation Cycling in COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Principal Investigator, BOUCHRA LAMIA, MD, PhD, University Hospital, Rouen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-A01690-47
Record Dates: First submitted 2015-10-29; First posted 2015-11-03 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: COPD
Keywords: COPD; Functional Electrical Stimulation Cycling; Pulmonary Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- One single arm group (Experimental): COPD included in a pulmonary rehabilitation program
  Intervention:
  Investigators used a bedside cycloergometer with electrical stimulation. COPD perform 2 measure of oxygen uptake during exercise for compare aerobic capacities:
  * Functional Electrical Stimulation Cycling (FES-cycling)
  * Classic Cycloergometer endurance training with a sham electrical stimulation
  Interventions: Device: FES-cycling; Device: Classic cycloergometer

INTERVENTIONS:
Device: FES-cycling — Patients performed an endurance tests with functional electrical stimulation during 30 minutes with an oxygen uptake measure.
Device: Classic cycloergometer — Patients performed an endurance tests on classic ergometer during 30 minutes with a sham electrical stimulation with an oxygen uptake measure.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) had systemic repercussion and lead to peripheral muscular dysfunction. Muscular atrophy limits aerobic capacity and is a major limitation of daily activity and quality of life. Technologies likes' neuromuscular electrical stimulation (NMES) are currently being adapted and tested to support exercise training.

The investigators hypothesized that functional electrical stimulation cycling improves VO2 and aerobic capacities during exercise compared to endurance training.

ELIGIBILITY:
Inclusion Criteria:

* COPD (Stade II, III or IV)
* Inform consent

Exclusion Criteria:

* Pulmonary rehabilitation contraindication
* Patient with Pacemaker
* Patient in acute exacerbation
* Patient with neurologic comorbidity
* Anemiae

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-04; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
oxygen uptake (VO2) | during 30 minutes exercise

SECONDARY OUTCOMES:
Ratio Ventilation/VO2 (Ventilation equivalent for oxygen) | during 30 minutes exercise
  Number of liters of air must be ventilated to consume 1 liter of O2
Ratio Ventilation/VCO2 (Ventilation equivalent for carbon dioxide) | during 30 minutes exercise
  Number of liters of air must be ventilated to reject 1 liter of CO2
cardiac output | during 30 minutes exercise
Muscular fatigue | after 30 minutes exercise

CONTACTS AND LOCATIONS:
Overall Officials: Clement Medrinal, Principal Investigator — Groupe Hospitalier du Havre
Locations (1):
- Medrinal, Montivilliers, France

REFERENCES:
- [Derived] Medrinal C, Prieur G, Combret Y, Quesada AR, Debeaumont D, Bonnevie T, Gravier FE, Dupuis Lozeron E, Quieffin J, Contal O, Lamia B. Functional Electrical Stimulation-A New Therapeutic Approach to Enhance Exercise Intensity in Chronic Obstructive Pulmonary Disease Patients: A Randomized, Controlled Crossover Trial. Arch Phys Med Rehabil. 2018 Aug;99(8):1454-1461. doi: 10.1016/j.apmr.2018.02.002. Epub 2018 Mar 7. PMID 29524398
- [Derived] Medrinal C, Prieur G, Debeaumont D, Robledo Quesada A, Combret Y, Quieffin J, Contal O, Lamia B. Comparison of oxygen uptake during cycle ergometry with and without functional electrical stimulation in patients with COPD: protocol for a randomised, single-blind, placebo-controlled, cross-over trial. BMJ Open Respir Res. 2016 Apr 12;3(1):e000130. doi: 10.1136/bmjresp-2016-000130. eCollection 2016. PMID 27110364